CLINICAL TRIAL: NCT02909166
Title: Role of ALiskiren, a Direct Renin Inhibitor, in Preventing Atrial Fibrillation in Patients With a Pacemaker; RALF. A Double-blind, Randomized, Parallel-group, Single Centre Study
Brief Title: Role of ALiskiren, a Direct Renin Inhibitor, in Preventing Atrial Fibrillation in Patients With a Pacemaker; RALF.
Acronym: RALF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mika Lehto (Other)
Responsible Party: Sponsor-Investigator, Mika Lehto, MD, PhD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RALF
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aliskiren (Active Comparator): Aliskiren 300 once a day (q.d)
  Interventions: Drug: aliskiren
- placebo (Placebo Comparator): Placebo once a day (q.d)
  Interventions: Drug: aliskiren

INTERVENTIONS:
Drug: aliskiren
  Other Names: Rasilez

SUMMARY:
The aim of the study is to find out whether aliskiren reduces atrial fibrillation burden measured with a pacemaker device

DETAILED DESCRIPTION:
The aim of the study is to find out the effect of a direct renin inhibitor, aliskiren, in reduction of AF with patients who have a pacemaker due to sinus node disease and paroxysmal atrial fibrillation.

Hypothesis is that there is a possibility to reduce atrial remodeling due to AF and also to enhance atrial reverse remodeling with aliskiren. The effect of aliskiren to total AF burden will be evaluated from the pacemaker's memory storage.

The main purpose of the study is to find new and safe drug treatments targeting to reduce AF recurrences and related complications in pacemaker patients. Also the aim is to evaluate the feasibility of a modern and highly sophisticated pacemaker system in the evaluation of drug treatment with AF reduction.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 85 years
* sinus node disease and paroxysmal AF
* provided signed informed consent according to the Declaration of Helsinki for study participation
* a previously implanted St. Jude Medical Identity / Victory / Zephyr ADX or any newer model of SJM DDDR pacemaker with ability to record high atrial rates

Exclusion Criteria:

* contraindication for the use of aliskiren
* severe impairment of renal function (serum creatinine > 160 µmol/L) or patient with solitary kidney or renal transplant or renal artery stenosis
* significant known aortic or mitral valve stenosis or obstructive hypertrophic cardiomyopathy
* hypersensitivity to aliskiren or to any of the excipients
* concomitant treatment with cyclosporine
* patients with uncontrolled hypertension requiring treatment for hypertension
* systolic blood pressure measured in two separate occasions ≥ 160 mmHg
* diastolic blood pressure in two separate occasions ≥ 100 mmHg
* absolute indication for the use of an RAAS blocker
* chronic, persisting AF (persisting AF at screening with ≥ 4 cardioversions performed beforehand)
* sitting systolic arterial blood pressure of less than 100 mm Hg at the time of randomisation
* need for ventricular pacing more than 30% at the enrolment
* pregnancy and/or lactation
* women of childbearing potential (only postmenopausal women or women after tubal ligation will be allowed)
* other serious disease expected to cause substantial deterioration of patient's health during the next two years
* past or present alcohol or drug abuse
* participation in other clinical trials during the last three months
* suspicion of poor study compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
burden of atrial fibrillation | From the start of the study to the end of the study; 0 - 12 months

SECONDARY OUTCOMES:
number of AF episodes | From the start of the study to the end of the study; 0 - 12 months
number of persistent AF episodes lasting more than 48 hours | From the start of the study to the end of the study; 0 - 12 months
the length of the paced P-wave measured by high resolution ECG (SAECG) | after each 6-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No